CLINICAL TRIAL: NCT01058122
Title: Collection, Evaluation and Assessment of Adverse Drug Reactions on the Oncology Ward
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Marco Egbring, MD, University of Zurich
Other Study IDs: kein Sponsor
Record Dates: First submitted 2009-12-15; First posted 2010-01-28 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Adverse Drug Reactions
Keywords: Adverse drug reactions in patients on the oncology ward
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients on the ward
  Interventions: Procedure: Collection of adverse drug events

INTERVENTIONS:
Procedure: Collection of adverse drug events

SUMMARY:
The proposed cohort study collected within a 5-month observation period adverse drug reaction (Adverse Drug Events - ADE) in patients at the Department of Oncology at the University of Zurich. ADE have been recorded using prospective monitoring and assessed using standardized algorithms regarding causality and severity. Data sources included information from the medical records, laboratory values and internal rounds. Additional information has been collected using a standardized patient questionnaire.

The primary endpoints of this study are to determine the frequency of ADE, the comparison of the quality of data sources and collection methods for the detection of ADE in regard to patient characteristics, size, number of medications, the category of ADE, severity, causation, diagnosis, hospitalization, cause of hospitalization and medication cause. Secondary endpoint is the assessment of the ADE causality, severity and predictability.

ELIGIBILITY:
Inclusion criteria:

* German-speaking patients,
* At least 18 years old.

Exclusion criteria:

* Patients who could not give her consent, or have given, and any minor patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized at the oncology ward G and H of the university hospital zurich during the 5-month observation period
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University hospital zurich, Zurich, Canton of Zurich, Switzerland